CLINICAL TRIAL: NCT07099833
Title: Aetiology and Pattern of Mandibular Condylar Fractures: A Retrospective Cohort Study of 122 Patients
Brief Title: Aetiology and Pattern of 122 Patients With Mandibular Condylar Fracture
Status: Completed | Type: Observational
Sponsor: Azita Sadeghzade (Other)
Responsible Party: Sponsor-Investigator, Azita Sadeghzade, Assistant Professor of Oral and Maxillofacial Medicine, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Other Study IDs: IR.SUMS.DENTAL.REC.1399.120
Record Dates: First submitted 2025-06-27; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Mandibular Fractures; Facial Injuries
Keywords: Mandibular Condylar Fracture; Subcondylar Fracture; Craniofacial Trauma
MeSH Terms: conditions — Mandibular Fractures; Facial Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 100 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Azita Sadeghzade — Azita Sadeghzade

SUMMARY:
This retrospective observational study aimed to investigate the aetiology and fracture patterns among patients with mandibular condylar fractures (MCF) who were treated at a trauma center in Shiraz, Iran, between 2018 and 2020. A total of 122 patients were included. The study involved collecting data on fracture characteristics, including anatomical location, classification (MacLennan and Loukota systems), angle of fracture lines, and the presence of concomitant maxillofacial injuries. The objective was to examine correlations between these characteristics and demographic or clinical factors such as age, sex, and mechanism of injury.

DETAILED DESCRIPTION:
This is a retrospective cohort study conducted at a major trauma center affiliated with Shiraz University of Medical Sciences, Iran. The study enrolled patients diagnosed with unilateral or bilateral mandibular condylar fractures between January 2018 and December 2020. Data were extracted from clinical records and radiographic evaluations. Fractures were classified according to the MacLennan and Loukota systems, and relevant demographic and injury-related information was recorded. No interventions were administered as part of this registry. All procedures were conducted under approval from the institutional ethics committee. The primary aim was to investigate patterns in fracture characteristics and their associations with trauma mechanisms and patient demographics.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral or bilateral mandibular condylar fracture
* Trauma-related fracture confirmed by clinical and radiographic evaluation
* Complete medical record and imaging data available
* Age between 12 and 65 years at the time of trauma

Exclusion Criteria:

* History of prior mandibular condylar fracture
* Incomplete medical or imaging records
* Patients younger than 12 or older than 65 at time of injury

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 12 to 65 years with trauma-induced unilateral or bilateral mandibular condylar fractures who were admitted to a trauma center affiliated with Shiraz University of Medical Sciences between January 2018 and December 2020. All included patients had complete clinical and radiographic records and no prior history of condylar fracture.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Distribution of mandibular condylar fracture types (MacLennan classification) | At initial evaluation (2018-2020)
  Frequency and percentage of fracture types (Class I-IV) based on MacLennan classification at initial clinical evaluation.
Anatomical location of mandibular condylar fractures | At initial evaluation (2018-2020)
  Distribution of fracture sites: subcondylar, condylar neck, or condylar head based on CT scan classification (Loukota system).
Etiology of mandibular condylar fractures | At initial evaluation (2018-2020)
  Proportion of fractures attributed to road traffic accident, falling, or assault based on patient report.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Sciences, Shiraz, Iran., Shiraz, Iran

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT07099833/Prot_000.pdf